CLINICAL TRIAL: NCT04168476
Title: Effectiveness of Scapula Mobilization Technique on Neural Mechanosensitivity of Upper Limb Neural Test 1 (ULNT1) in Subjects With Mechanical Neck Pain
Brief Title: Effectiveness of Scapula Mobilization on Mechanosensitivity of Upper Limb Neural Test 1 in Mechanical Neck Pain
Acronym: ULNT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aitor Vaquero Garrido (Other)
Responsible Party: Sponsor-Investigator, Aitor Vaquero Garrido, Research Master, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Upper Limb Neural Test 1
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Neck Pain; Musculoskeletal Diseases
Keywords: Median Nerve; Hand Strength; Brachial plexus; Physical Therapy Modalities; Neck Pain
MeSH Terms: conditions — Neck Pain; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized prospective controlled trial
Who Masked: Participant
Masking Description: Single-blind clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants of this group were assessed by the examiner twice, pre and post intervention, having recorded two values for each of the following variables:
  * Visual Analogue Scale
  * Range of movement
  * Hand grip strength. After a first assessment, scapula mobilization techniques were performed and participants reassessed.
  Interventions: Other: Interscapular muscle release or scapular mobilization technique as described by Travell and Simons.
- Control group (Placebo Comparator): Participants of this group were assessed by the examiner twice, pre and post intervention, having recorded two values for each of the following variables:
  * Visual Analogue Scale
  * Range of movement
  * Hand grip strength. The procedure was a contralateral calcaneus abduction and adduction mobilization technique was carried out.
  Interventions: Other: Calcaneus abduction and adduction mobilization technique

INTERVENTIONS:
Other: Interscapular muscle release or scapular mobilization technique as described by Travell and Simons. — Patient is sidelying with the testing side up. The auditor stands in front of the patient, reaches over the patient's shoulder to grasp the upper portion of the vertebral border of the scapula, and the other arm reaches under the patient's humerus to grasp the lower portion of the vertebral border of the scapula.
  The auditor then slowly moves the scapula into elevation/depression, internal/external rotation/abduction and adduction.
  To standardize the technique and be able to reproduce it in each participant, a set of 10 repetitions for each movement was performed in the same order.
  Arms: Treatment group
Other: Calcaneus abduction and adduction mobilization technique — Abduction and adduction mobilization of the calcaneus is carried out in the opposite side of the upper extremity measured.
  Arms: Control group

SUMMARY:
Between 45% and 70% of the general population suffers neck pain at some point in their lives, making it one of the most frequent reasons for taking sick leave. Given its importance in physiotherapy at clinical level, we seek to observe how a scapular mobilization technique might influence the neural mechanosensitivity of the median nerve as measured by Upper Limb Neural Test 1 (ULNT1) on subjects with neck pain.

Hypotheses and objectives. Performing a scapular mobilization technique on subjects with neck pain and a positive ULNT1 improves the patient's response to said test. It also decreases the patient's neck pain as measured using a Visual Analog Scale (VAS) for pain and increases grip strength.

Material and method. A single-blind clinical trial was performed on subjects randomly assigned to either a treatment group or control group. The sample consisted of 60 subjects (N = 60) -30 in the treatment group (n = 30) and the other 30 as a control (n = 30) -and was made up of patients with neck pain and a positive ULNT1. A scapular mobilization was performed on the first group and on the second, a calcaneus abduction adduction on the opposite side from the positive ULNT1 as a placebo.

DETAILED DESCRIPTION:
Mechanical cervicalgia is a very frequent and important clinical picture in physiotherapy consultations. It can be considered as a pluripatology as it covers somatic, functional, psychological and social aspects. This ailment is suffered by between 45 and 70% of the general population during some period of life and is one of the most frequent justifications of work leave and the main cause of permanent disability. Mechanical cervicalgia significantly decreases the quality of life of those who suffer from it: it frequently produces a significant disability when generating pain, functional deficit, headaches, movement restriction, vertiginous syndromes, nausea and / or vomiting, etc. This leads to reduced work time and increased health system costs, causing a strong economic and social impact. For example, Borghouts JA and Cols point out that in the Netherlands in 1996 these costs were approximately 686 million dollars, which constituted 1% of total health expenditure and 0.1% of its Gross Domestic Product (GDP) . In Spain, referrals to the cervicalgia physiotherapy service represent 10% of the total of all health demands; in Britain this percentage reaches 15% and in Canada 30%. Likewise, it should be considered that the direct cost caused by cervicalgia to the health system in our country, specifically to the Primary Care consultation, constitutes 2% of the total, and in some centers this figure reaches up to 12% if they are considered diagnostic tests, pharmaceutical expenses and visits to the specialist.

ELIGIBILITY:
Inclusion Criteria:

* Adults with mechanical cervicalgia and a positive median neurodynamic test (ULNT1) reproducing the patient's cervical pain.
* Sign the informed consent.

Exclusion Criteria:

* Do not sign informed consent.
* Patients who, due to previous malformations or injuries, are not able to be positioned in the position described for the ULNT1 test.
* Congenital malformations of the cervical spine and / or upper limb.
* Previous spine surgery.
* Neurological pathologies diagnosed, such as diabetic polyneuritis or others.
* Refusal to participate in the study.

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Goniometer Test | Two minutes
  The axis of the Goniometer is placed On the elbow joint. The stationary arm is lined up with the arm and the moveable arm along the forearm. The subject is asked to perform elbow extension and the angle is measured.
  Improvement of this angle 10º. Inmediately after the intervention

SECONDARY OUTCOMES:
Neck pain | Two minutes
  Improvement of this 0,5 Newtons. Using a visual pain scale, with values between 0 and 10, the subject marks the intensity level of the neck pain. Inmediately after the intervention

OTHER OUTCOMES:
Hand pressing force | Five minutes
  To measure the grip force of the hand we use the Dynamometer hydraulic baseline (SP-5030J1). We always place the subject in the same position to ensure that the conditions were the same, seated subject, shoulder adducted and in neutral rotation, 90º bend of the elbow, neutral position of the forearm, wrist in slight dorsal flexion (always between 0º and 30º) and a cubital deviation between 0º and 15º.

CONTACTS AND LOCATIONS:
Overall Officials: Aitor Vaquero Garrido, Study Chair — University of Seville
Locations (1):
- Aitor Vaquero Garrido, Seville, Spain

IPD SHARING:
Plan to Share IPD: No